CLINICAL TRIAL: NCT04697147
Title: Rescuing Neurodevelopment in Zika-Exposed Infants in Grenada
Brief Title: Zika and Neurodevelopment Among Infants in Grenada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Windward Islands Research and Education Foundation (Other)
Collaborators: St. George's University (Unknown); Stanford University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dr. Randall Waechter, Associate Director of Research, Windward Islands Research and Education Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGUZIKV
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Zika Virus Infection; Neurocognitive Deficit; Development, Child; Neurodevelopmental Abnormality
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neurocognitive assessors are blinded to which participants have received the intervention during their longitudinal visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Immediately randomized to receive the intervention for 12 weeks.
  Interventions: Behavioral: Conscious Discipline-Based Environmental Enrichment Intervention
- Waitlist Control (No Intervention): Randomized to receive the intervention post-study.

INTERVENTIONS:
Behavioral: Conscious Discipline-Based Environmental Enrichment Intervention — Conscious Discipline, a social-emotional skills-based learning program that draws on current brain research and fosters enhanced connections between parents and their children.
  Arms: Intervention Group

SUMMARY:
Implement a randomized controlled trial, evidence-based, culturally adapted, environmental enrichment intervention for the purpose of enhancing neurocognitive outcomes among Zika Exposed Children.

DETAILED DESCRIPTION:
The intervention group received up to twelve 1-hour weekly visits by trained and experienced Grenadian parent and infant relationship specialists who provided home-based interventions as part of the Saving Brains Grenada project.

The environmental enrichment intervention is a brain-based program that teaches parents about brain development in young infants and skills for building a strong social-emotional connection that stimulates brain development and maximizes neurocognitive function. A detailed intervention manual was developed and used as a guide for the intervention specialists. Neurocognitive outcomes in the intervention and control group were assessed pre and post intervention by a separate and blinded assessment team.

ELIGIBILITY:
Inclusion Criteria:

* Must be actively enrolled in the pre-existing Zika Cohort Study
* Infant must be alive and living with a parent/guardian at the time of recruitment
* Infant must be between 24-27 months at the time of recruitment

Exclusion Criteria:

* Any infants older than 27 months
* Persons not enrolled in the pre-existing Zika Cohort Study

Ages: 24 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The INTERGROWTH 21st Neurodevelopmental Assessment (INTER-NDA) | 22-30 months
  The INTER-NDA is a measure of cognition, motor skills (fine and gross motor), language (expressive and receptive), behavior, executive function, attention and social-emotional reactivity for 2-year-olds. The measure is comprised of 30 items scored across a spectrum, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Waechter, PhD, Principal Investigator — Windward Islands Research and Education Foundation
Locations (1):
- Windward Islands Research and Education Foundation (WINDREF), Saint George's, Grenada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waechter R, Burgen KS, Punch B, Evans R, Blackmon K, Noel T, Fernandes M, Landon B. Improving neurodevelopment in Zika-exposed children: A randomized controlled trial. PLoS Negl Trop Dis. 2022 Mar 8;16(3):e0010263. doi: 10.1371/journal.pntd.0010263. eCollection 2022 Mar. PMID 35259172